CLINICAL TRIAL: NCT04410575
Title: Mental Health Assessment and Prescribing by Alberta Pharmacists (MAP-AP)
Brief Title: Mental Health Assessment and Prescribing by Alberta Pharmacists
Acronym: MAP-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB ID Pro00093776
Record Dates: First submitted 2020-05-21; First posted 2020-06-01 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder; Pharmacist-Patient Relations
Keywords: Pharmacist; Prescribing; Major Depressive Disorder; Generalized Anxiety Disorder; Mental Health; Intervention; Expanded Scope
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Psychological Well-Being | interventions — Deprescriptions

STUDY DESIGN:
Intervention Model Description: Multi-center randomized control trial evaluating the mean difference in depression and anxiety score with patients with major depressive disorder (MDD) and/or generalized anxiety disorder (GAD) by pharmacists with prescribing & management interventions in comparison to pharmacist management per standard pharmacist care.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Stratified randomization of participants via blocking factor to either pharmacist intervention or standard pharmacist care groups.
  Participants will be assigned a unique identifier number & group allocation for the duration of their participation in the study (also recorded by the pharmacy partner to ensure consistency in the delivery of pharmacist interventions described by the participant's group allocation.
  The participant is sent a secured electronic link (to the contact number or email they provided in the written consent form) of the electronic version of the PHQ-9/GAD-7 questionnaire tool to complete.
  The study data (from the participant's electronic questionnaire tool results) will be sent directly to a centralized & secured website/spreadsheet to ensure allocation concealment for the investigational team. The participant will report their score to the pharmacist participant through an electronic recording platform
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Standard Pharmacist Care + Pharmacist Interventions) (Experimental): Participants enrolled in the intervention group will receive pharmacist interventions, in addition to standard care (as outlined in the Alberta College of Pharmacist Standards of Practice for Pharmacist and Pharmacy technicians), at enrollment (month 0) and at 1, 3, and 6 month in-person follow-up appointments
  Interventions: Other: Standard Pharmacist Care; Other: Reviewed Questionnaire tool results with participant; Other: Patient Clinical Assessment; Other: Psychotherapy Referral; Other: Pharmacist initiated interim telephone follow-up with participant; Other: Communication update with physician after participant contact; Other: Medication Counselling and Educational Support; Other: Non-medication Counselling; Other: Identification of drug interaction; Other: Identification of drug adverse effect; Other: Identification of severe deterioration; Other: Pharmacist-to-physician recommendation for medication adjustment, change to alternative, add-on, or deprescribing; Other: Pharmacist initiated medication adjustment, change to alternative, add-on, or deprescribing
- Control Group (Standard Pharmacist Care) (Active Comparator): Patients randomized to the usual care group will receive standard pharmacy care (as outlined in the Alberta College of Pharmacist Standards of Practice for Pharmacist and Pharmacy technicians) and physician care, at enrollment (month 0) with no specific interventions for the duration of 6 months, until the 6 month in-person follow-up appointment
  Interventions: Other: Standard Pharmacist Care; Other: Medication Counselling and Educational Support; Other: Non-medication Counselling; Other: Identification of drug interaction; Other: Identification of drug adverse effect; Other: Identification of severe deterioration; Other: Pharmacist-to-physician recommendation for medication adjustment, change to alternative, add-on, or deprescribing

INTERVENTIONS:
Other: Standard Pharmacist Care — Standard pharmacy care (as outlined in the Alberta College of Pharmacist Standards of Practice for Pharmacist and Pharmacy technicians)
Other: Reviewed Questionnaire tool results with participant — Pharmacist reviews results of the patient-administered PHQ-9 and/or GAD-7 questionnaire tool, at the scheduled follow-up appointment
  Arms: Intervention Group (Standard Pharmacist Care + Pharmacist Interventions)
Other: Patient Clinical Assessment — Pharmacist conducts clinical assessment of the participant's major depressive disorder and/or generalized anxiety, which can include: appearance, current mood, sleeping patterns, mental health, medical history, social history, family history, relationship with others, suicidal ideation, previous suicide attempts or hospitalizations, current employment status
  Arms: Intervention Group (Standard Pharmacist Care + Pharmacist Interventions)
Other: Psychotherapy Referral — Pharmacist initiates collaboration with physician to arrange referral for psychotherapy, including: psychologist, social worker, counsellor, psychiatrist
  Arms: Intervention Group (Standard Pharmacist Care + Pharmacist Interventions)
Other: Pharmacist initiated interim telephone follow-up with participant — Interim telephone follow-up conducted by the pharmacist since the last in-person follow-up & a minimum of 1-2 weeks after the last in-person follow-up that involved a dose adjustment, prescribing of adjunctive medication, or discontinuation of therapy (Note: a telephone follow-up does not replace the scheduled in-person follow-up)
  Arms: Intervention Group (Standard Pharmacist Care + Pharmacist Interventions)
Other: Communication update with physician after participant contact — Pharmacist provides communication update (fax or electronic charting) with the participant's physician after contact with the participant
  Arms: Intervention Group (Standard Pharmacist Care + Pharmacist Interventions)
Other: Medication Counselling and Educational Support — Pharmacist provides medication related counselling and educational support to participant
Other: Non-medication Counselling — Pharmacist provides non-medication related counselling and educational support to participant
Other: Identification of drug interaction — Pharmacist identification of drug interaction related to medication for major depressive disorder and/or generalized anxiety
Other: Identification of drug adverse effect — Pharmacist identification of adverse effect related to medication for major depressive disorder and/or generalized anxiety
Other: Identification of severe deterioration — Pharmacist identification of participant severe deterioration (i.e. suicide attempt)
Other: Pharmacist-to-physician recommendation for medication adjustment, change to alternative, add-on, or deprescribing — Pharmacist collaborates, discusses, and makes recommendations to physician re: treatment plan for MDD and/or GAD (as per CANMAT guidelines), which can include: medication dose adjustment, change to alternative medication, add-on, or deprescribing
Other: Pharmacist initiated medication adjustment, change to alternative, add-on, or deprescribing — Pharmacist initiated alteration to treatment plan for MDD and/or GAD (as per CANMAT guidelines), which can include: medication dose adjustment, change to alternative medication, add-on, or deprescribing
  Arms: Intervention Group (Standard Pharmacist Care + Pharmacist Interventions)

SUMMARY:
This is a clinical trial evaluating the experimental intervention of enhanced pharmacist care by pharmacists with additional prescribing authorization (APA) in Alberta, for patients newly diagnosed with Major Depressive Disorder (MDD) and Generalized Anxiety Disorder (GAD).

DETAILED DESCRIPTION:
Primary objective

-To evaluate the effect of enhanced pharmacist care possible by community pharmacists with APA in comparison with usual care (standard pharmacist care and physician care) for patients with MDD and/or GAD initiated on pharmacotherapy, with focus on interventions that include:

i) monitoring (lab ordering and interpretation, clinical monitoring of MDD and GAD) ii) patient education iii) referral facilitation (in collaboration with prescribing physician) iv) prescribing (dose adjustment and the addition of adjunctive medication)

Secondary objectives

* To evaluate the effect of APA pharmacist interventions on:

  i)Clinical:
* The rate of achieving clinical response and remission of MDD and/or GAD compared to usual care (using PHQ-9/GAD-7)
* Change in the mean PHQ-9 and GAD-7 score
* Cognitive and functional impairment related to MDD and/or GAD
* The occurrence of relapse of depression and/or anxiety
* The proportion of patients receiving appropriate and optimized depression and anxiety medication
* Patient complaints and/or experiences of medication-related side effects during treatment for MDD and/or GAD (i.e. GI intolerance, dizziness, weight gain)

ii) Process:

* The impact of the interventions on patient satisfaction and quality of life impact (Patient survey)
* Assure sustainability by exploring enabling (i.e. pharmacist reimbursement framework) and potential barrier forces (i.e. pharmacist training in managing patients with MDD and GAD)

ELIGIBILITY:
Inclusion criteria:

* Adults (≥ 18 years of age) newly diagnosed with MDD and/or GAD, including:
* Patients starting on medications for the management of adults with MDD
* Patients starting on medications for the management of GAD

Exclusion Criteria:

* Pregnancy
* Non-Alberta residents
* Unwilling or unable to participate in regular follow-up visits
* Unwilling to participate/sign consent form
* ≥2 suicide attempts per year
* Severe, psychotic, and catatonic depression
* History of and/or current substance abuse, intoxication, addiction or withdrawal
* Patients diagnosed with comorbid anxiety disorders other than GAD, including: panic -disorder, agoraphobia, specific phobia, social anxiety disorder, obsessive-compulsive disorder, posttraumatic stress disorder
* Patients diagnosed with comorbid depressive disorder other than MDD, including: depressive disorder due to another medical condition (e.g. hypothyroidism, MS, OSA, -Parkinsons, stroke, TBI, Vitamin B12 insufficiency, Huntington disease, adrenal insufficiency, mononucleosis, systemic lupus erythematosus), adjustment disorder with depressed mood
* Patients diagnosed with concurrent ADHD, bipolar disorder, schizophrenia and schizoaffective disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Mean score difference in Patient Health Questionnaire 9-item (PHQ-9) score | 6 months
  Mean score difference in PHQ-9 score from baseline to end of study between intervention (pharmacist intervention + standard pharmacist care) group vs control (standard pharmacist care) group;
  PHQ-9 scores reflect depression severity, ranges from 0-27 (Scores: 0-4 none/minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe)
Mean score difference in Generalized Anxiety Disorder 7-item (GAD-7) score | 6 months
  Mean score difference in GAD-7 score from baseline to end of study between intervention (pharmacist intervention + standard pharmacist care) group vs control (standard pharmacist care) group;
  GAD-7 scores reflect anxiety severity; Ranges from 0-21 (Scores: 0-4 none/minimal. 5-9 mild, 10-14 moderate, 15-21 severe)

SECONDARY OUTCOMES:
Difference in proportion of participants achieving clinically significant treatment response in Patient Health Questionnaire 9-item (PHQ-9) score between pharmacist intervention vs. standard pharmacist care | 6 months
  Clinically significant treatment response for the PHQ-9 is defined as a reduction in PHQ-9 score by at least 50% from baseline;
  PHQ-9 Scores reflect depression severity, ranges from 0-27 (Scores: 0-4 none/minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe)
Difference in proportion of participants achieving clinically significant treatment response in Generalized Anxiety Disorder 7-item (GAD-7) score between pharmacist intervention vs. standard pharmacist care | 6 months
  Clinically significant treatment response for the GAD-7 is defined as a reduction in GAD-7 score by at least 50% from baseline;
  GAD-7 scores reflect anxiety severity; Ranges from 0-21 (Scores: 0-4 none/minimal. 5-9 mild, 10-14 moderate, 15-21 severe)
Difference in the proportion of participants with Major Depressive Disorder (MDD) to achieve Patient Health Questionnaire 9-item (PHQ-9) score <5 | 6 months
  Difference in the proportion of participants with MDD to achieve PHQ-9 score <5 (i.e. remission/no depression) between the pharmacist intervention and standard pharmacist care groups
  PHQ-9 scores reflect depression severity; Ranges from 0-27 (Scores: 0-4 none/minimal, 5-9 mild, 10-14 moderate, 15-19 moderately severe, 20-27 severe)
Difference in the proportion of participants with Generalized Anxiety Disorder (GAD) to achieve Generalized Anxiety Disorder 7-item (GAD-7) score <5 | 6 months
  Difference in the proportion of participants with GAD to achieve GAD-7 score <5 (i.e. remission/no anxiety) between the pharmacist intervention and standard pharmacist care groups;
  GAD-7 scores reflect anxiety severity; Ranges from 0-21 (Scores: 0-4 none/minimal. 5-9 mild, 10-14 moderate, 15-21 severe)
Percentage difference in self-reported safety concerns disclosed by participant to pharmacist partner, between intervention (pharmacist intervention + standard pharmacist care) and control (standard pharmacist care) study groups, during the study period. | 6 months
  The participant discloses to the pharmacist partner at any time during the duration of study, events that fit the description of a safety concern and measured via frequency of occurrence.
  Safety concerns include:
  1) Adverse Medication Effects 2) Suicide Ideation/attempt, 3) Causing withdrawal from Study

CONTACTS AND LOCATIONS:
Overall Officials: Yazid Al Hamarneh, BSc (Pharm), PhD, CDM, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No